CLINICAL TRIAL: NCT07184749
Title: Neurocognitive and Psychological Impact of Chemotherapy in Breast Cancer Patients: A Prospective Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alshaymaa Abdelghaffar, Assistant Professor, Sohag University
Other Study IDs: Soh-Med-25-7-8PD; Sohag University (Other: Sohag University)
Record Dates: First submitted 2025-08-30; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Despite growing awareness of neurocognitive and psychological complications of systemic chemotherapy administration in breast cancer, prospective observational studies evaluating such effects in Egyptian breast cancer patients-especially with pre- and post-treatment assessments-remain limited. Given the rising incidence of breast cancer in Egypt and the growing population of long-term survivors, it is essential to investigate the extent and nature of cognitive and psychological changes associated with treatment. The current study aims to fill this gap by prospectively evaluating neurological, cognitive, and psychological parameters in newly diagnosed breast cancer patients, using validated tools before and one year after treatment.

DETAILED DESCRIPTION:
Patient Recruitment This prospective observational study will include female breast cancer patients who will be recruited from the neuropsychiatry, Clinical Oncology, and general surgery departments, as well as from outpatient clinics at Sohag University Hospital.

Inclusion Criteria Female patients with newly diagnosed breast cancer will be included. All patients will be evaluated before the initiation of treatment and again one year after treatment completion.

Study Methodology

All enrolled patients will undergo the following assessments:

Complete History taking: thorough medical, neurological, and oncological history will be obtained, including comorbidities and current medications.

Neurological Examination: Each patient will receive a comprehensive clinical neurological examination at baseline and one year after treatment.

Neuroimaging: Brain MRI will be performed to detect any structural brain abnormalities or metastatic lesions.

Neurophysiological Assessment Nerve conduction studies (NCS) will be conducted to evaluate for peripheral neuropathy.

Cognitive Function Assessment

Cognitive testing will be carried out at baseline and at the one-year follow-up using the following tools:

A. Wisconsin Card Sorting Test (WCST) This test will assess executive functions such as cognitive flexibility and set shifting.

Higher perseverative error scores will indicate poorer performance (7). B. Trail Making Test (TMT), Parts A & B Part A: Patients will connect sequential numbers to assess visual attention and processing speed.

Part B: Patients will alternate between numbers and letters (1-A-2-B…) to assess executive functioning.

Errors will be corrected by the examiner in real time (8). C. Montreal Cognitive Assessment (MoCA) This test will evaluate attention, memory, language, executive functions, visuospatial skills, and orientation.

Total score: 0-30, with higher scores indicating better function. (Nasreddine et al., 2005)

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed breast cancer female patients.
2. Chemotherapy is indicated for these patients either preoperative or postoperative.

Exclusion Criteria:

1. known history of neurological disease.
2. presence of symptoms suggesting positive neurological disease.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with newly diagnosed breast cancer for whom chemotherapy is prescribed
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
chemotherapy-induced peripheral neuropathy | 1 year, 2 years
  FACT/GOG-Ntx questionnaire
psychological impact of chemotherapy adminstration | 1 year, 2 years
  Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) questionnaire
  Total Neuropathy Score (TNS)
  EORTC QLQ-CIPN20 questionnaire
  Patient Neurotoxicity Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alshaymaa Ahmed, MD, PhD, Principal Investigator — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt